CLINICAL TRIAL: NCT00990028
Title: Effect of Rosuvastatin on Immunological Markers After Traumatic Brain Injury: Clinical Randomized Double Blind Study Phase 2
Brief Title: Effect of Rosuvastatin on Cytokines After Traumatic Brain Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other); AstraZeneca (Industry)
Responsible Party: Dr. Martin Sanchez, Clinical Epidemiology UASLP
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 28-09ROHI
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Head Injury
Keywords: moderate head injury; rosuvastatin; statin; amnesia; orientation
MeSH Terms: conditions — Craniocerebral Trauma; Amnesia; Orientation, Spatial | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental): 20 mg oral during 10 days
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg oral, for 10 days
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — 20 mg vehicle
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether rosuvastatin could alter the immunological response after head injury by modulating TNF-alpha,IL6,IL-1.

DETAILED DESCRIPTION:
The head injury is a frequent problem of health, which produces high morbid-mortality. Today is the main cause of death and disability between 18 and 40 years. In addition it originates expensive expenses in health care systems.

Head injury produces damage by primary mechanisms related to impact, then by biochemical ways which are activated and they carry to secondary damage. Many studies have been conducted for explaining secondary injury, the majority conclude there is a kind of ischemic lesion related maybe with changes in cerebral flow and metabolism. All these changes are associated to a immunological response. Up to now some drugs are directed to modulate the immunological system, although many of them have been ineffective.

Statins o inhibitors of HMG CoA reductase are drugs used in dyslipidemia, frequently for reduction in LDL. Experimental and clinical studies in stroke have shown improvement in outcome. The toxicity related to statin is myopathy and hepatopathy, both with low incidence without fatal cases. Rosuvastatin has been postulated be the most powerful with longest life and toxicity similar to another statins. Many studies have suggested an important immunomodulator effect after statins administration, The investigators have previously demonstrated the possible effect of statin on amnesia and disorientation improvement with patients who suffered a moderated head injury (Glasgow 9-13). The aim of this new study is to analyze the possible immunomodulator role of statins on head injury.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 16 and < 60 years old with HI less 24 hours in progression and Glasgow between < 13
* Acceptance of family to participate (first grade)

Exclusion Criteria:

* Previous head injury with severe disability
* History of neurological or psychiatric disease with severe disability
* Administration 24 hrs previous of: fibrates, niacin, ciclosporin, azoles, macrolides, inhibitors of protease, nefazodone, verapamil, diltiazem,amiodarone
* Very poor possibilities for survival
* Use of Administration of THAM, mannitol, barbiturates, corticosteroids, scavengers of free radicals, inhibitors of lipidic peroxidation, indometacin, calcium antagonist, antagonists of neurotransmitters before randomization
* isolated lesions in brain stem
* Allergy to the drug
* Hepatopathy or myopathy (or) history of this, or clinical data of hepatic disease
* Management previous in other Hospital
* Pregnancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasmatic levels of cytokines (IL-1B, IL-6, TNF-alfa) (pg/dL) | Day 3

SECONDARY OUTCOMES:
Functional outcome by Disability Rating Scale | after 3 months
change of lesions on CT scan | 72 hours
Determination of CK, AST, ALT | 3rd and 7th day
Amnesia time using GOAT Score | in-patient follow-up, after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gordillo-Moscoso, PhD, Study Chair — Clinical Epidemiology UASLP; Martin Sanchez-Aguilar, MSc, Principal Investigator — Clinical epidemiology UASLP
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Tapia-Perez H, Sanchez-Aguilar M, Torres-Corzo J, Rodriguez-Leyva I, Herrera-Gonzalez LB. [Statins and brain protection mechanisms]. Rev Neurol. 2007 Sep 16-30;45(6):359-64. Spanish. PMID 17899518
- [Background] Tapia-Perez J, Sanchez-Aguilar M, Torres-Corzo JG, Gordillo-Moscoso A, Martinez-Perez P, Madeville P, de la Cruz-Mendoza E, Chalita-Williams J. Effect of rosuvastatin on amnesia and disorientation after traumatic brain injury (NCT003229758). J Neurotrauma. 2008 Aug;25(8):1011-7. doi: 10.1089/neu.2008.0554. PMID 18690806
- [Background] Tapia-Perez H, Sanchez-Aguilar M, Torres-Corzo JG, Rodriguez-Leyva I, Gonzalez-Aguirre D, Gordillo-Moscoso A, Chalita-Williams C. Use of statins for the treatment of spontaneous intracerebral hemorrhage: results of a pilot study. Cent Eur Neurosurg. 2009 Feb;70(1):15-20. doi: 10.1055/s-0028-1082064. Epub 2009 Feb 5. PMID 19197830
- [Background] Tapia-Perez JH, Sanchez-Aguilar M, Schneider T. The role of statins in neurosurgery. Neurosurg Rev. 2010 Jul;33(3):259-70; discussion 270. doi: 10.1007/s10143-010-0259-4. Epub 2010 Apr 29. PMID 20429022
- [Derived] Sanchez-Aguilar M, Tapia-Perez JH, Sanchez-Rodriguez JJ, Vinas-Rios JM, Martinez-Perez P, de la Cruz-Mendoza E, Sanchez-Reyna M, Torres-Corzo JG, Gordillo-Moscoso A. Effect of rosuvastatin on cytokines after traumatic head injury. J Neurosurg. 2013 Mar;118(3):669-75. doi: 10.3171/2012.12.JNS121084. Epub 2013 Jan 4. PMID 23289819